CLINICAL TRIAL: NCT01999075
Title: Stacking Exercises Attenuate the Decline in Forced Vital Capacity and Sick Time (STEADFAST)
Brief Title: Stacking Exercises Aid the Decline in FVC and Sick Time
Acronym: STEADFAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Jesse's Journey (Other)
Responsible Party: Principal Investigator, Sherri Katz, Dr. Sherri Katz, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12/26E
Record Dates: First submitted 2013-11-14; First posted 2013-12-03 (Estimated); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Pulmonary complications; Lung volume recruitment,; Breath-stacking,; Cough efficacy,; Maximal insufflation capacity
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Treatment (Placebo Comparator): Conventional Treatment
  Interventions: Other: Conventional Treatment
- Lung Volume Recruitment (Active Comparator): Conventional treatment plus the use of Lung Volume Recruitment (LVR) twice per day
  Interventions: Device: Lung Volume Recruitment (LVR); Other: Conventional Treatment

INTERVENTIONS:
Device: Lung Volume Recruitment (LVR) — LVR will be used twice per day
  Arms: Lung Volume Recruitment
Other: Conventional Treatment — This may include: a. Physiotherapy, consisting of percussion, active cycle of breathing and/or postural drainage; b. Nutritional support, consisting of oral or tube-fed dietary supplements; c. Antibiotics (oral or intravenous), if there is evidence of respiratory infection; d. Non-invasive positive pressure ventilation, if there is evidence of nocturnal hypoventilation or sleep-disordered breathing; e. Systemic steroids

SUMMARY:
Duchenne Muscular Dystrophy is complicated by weak breathing muscles and lung infections. "Lung volume recruitment" is a technique performed using a face mask or mouthpiece and a hand-held resuscitation bag to stack breaths, inflate the lungs and help clear the airways of secretions by increasing the forcefulness of a cough. We believe this will slow down the steady loss of lung function, prevent lung infection, and improve quality of life. Our aim is to compare the outcome of a group of individuals with DMD treated with standard care to another group that also receives lung volume recruitment. If effective, this study will change clinical practice by including twice-daily treatment as part of the standard of care for individuals with DMD, in order to improve their lung health and quality of life.

DETAILED DESCRIPTION:
Background: Respiratory complications are the primary cause of morbidity and mortality associated with childhood Duchenne Muscular Dystrophy (DMD). Involvement of the respiratory muscles leads to progressive hypoventilation and/or recurrent atelectasis and pneumonia secondary to decreased cough efficacy. Lung volume recruitment (LVR) is a means of stacking breaths to achieve maximal lung inflation (MIC), prevent micro-atelectasis, and improve cough efficacy. Although it has been recommended by some experts as the "standard of care" for individuals with neuromuscular disease, the strategy has not been widely implemented in DMD given the lack of clinical trials to date to support its efficacy as well as the additional burden of care required in a population already requiring multiple interventions.

Primary Objective: To determine whether LVR, in addition to conventional treatment, is successful in reducing decline from baseline in forced vital capacity (FVC) over 2 years (percent predicted, measured according to American Thoracic Society standards), compared to conventional treatment alone in children with DMD.

Secondary Objectives: To determine differences between children treated with LVR in addition to conventional treatment, compared to those treated with conventional treatment alone, in: (1) the number of courses of antibiotics, hospitalizations and intensive care admissions for respiratory exacerbations, (2) health-related quality of life, and (3) peak cough flow and other pulmonary function tests.

Methods: We propose a 3-year multi-centre randomized controlled trial involving fifteen tertiary care pediatric hospitals across Canada. The study population consists of boys aged 6-16 years with DMD and FVC ≥ 30% of predicted. A sample size of 110 participants will be enrolled. This has been informed by chart review and survey of participating centres to be feasible, and will be re-assessed with an ongoing internal pilot study. Intervention: Participants will be allocated with a minimization procedure to receive conventional treatment (non-invasive ventilation, nutritional supplementation, physiotherapy and/or antibiotics, as decided by the treating physician) or conventional treatment plus twice daily LVR exercises performed with an inexpensive, portable self-inflating resuscitation bag containing a one-way valve and a mouthpiece. Data Analysis: The primary outcome (change in percent predicted FVC over 2 years) will be compared between the two study groups using an analysis of co-variance (ANCOVA) that takes into account baseline FVC and minimization factors.

Importance: Decline in pulmonary function among children with DMD negatively affects quality of life and predicts mortality. The relatively simple strategy of LVR has the potential to optimize pulmonary function and reduce respiratory exacerbations, thereby improving quality of life for individuals with DMD. This study is novel in that it is the first randomized controlled trial of LVR. A major strength is that the results will give support or refute recommendations regarding inclusion of LVR in the standard of care for individuals with DMD worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-16 years - This age range was selected as there are accepted normative pulmonary function data and children 6 years of age and older are generally able to reliably perform pulmonary function tests. Children are followed in participating centres until they reach 18 years of age (allowing two years of follow-up).
* Clinical phenotypic features consistent with DMD and confirmed by either: (1) Muscle biopsy showing complete dystrophin deficiency; (2) Genetic test positive for deletion or duplication in the dystrophin gene resulting in an 'out-of-frame' mutation; or (3) Dystrophin gene sequencing showing a mutation associated with DMD.
* FVC ≥ 30% predicted - This range of pulmonary function was selected to exclude those with severe restrictive respiratory impairment, who are less likely to be able to reliably perform pulmonary function testing over a two year period.
* A caregiver willing to provide the therapy
* Fluency in English or French

Exclusion Criteria:

* Unable to perform pulmonary function tests and/or LVR manoeuvre
* Presence of an endotracheal or tracheostomy tube
* Already using LVR and/or the Respironics in-exsufflator between and during respiratory infections
* Known susceptibility to pneumothorax or pneumomediastinum
* Uncontrolled asthma or other obstructive lung disease
* Symptomatic cardiomyopathy (ejection fraction less than 50% )

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2013-03; Primary Completion 2018-11-22 (Actual); Study Completion 2018-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherri Katz, MD, Principal Investigator — Children's Hospital of Eastern Ontario; Ian MacLusky, MD, Study Director — Children's Hospital of Eastern Ontario; Nicholas Barrowman, PhD, Study Director — Children's Hospital of Eastern Ontario
Locations (9):
- Canada (9):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario
  - London Health Sciences, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario
  - SickKids Hospital, Toronto, Ontario
  - Hôpital Ste. Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Katz SL, Mah JK, McMillan HJ, Campbell C, Bijelic V, Barrowman N, Momoli F, Blinder H, Aaron SD, McAdam LC, Nguyen TTD, Tarnopolsky M, Wensley DF, Zielinski D, Rose L, Sheers N, Berlowitz DJ, Wolfe L, McKim D. Routine lung volume recruitment in boys with Duchenne muscular dystrophy: a randomised clinical trial. Thorax. 2022 Aug;77(8):805-811. doi: 10.1136/thoraxjnl-2021-218196. Epub 2022 Mar 2. PMID 35236763
- [Derived] Morrow B, Argent A, Zampoli M, Human A, Corten L, Toussaint M. Cough augmentation techniques for people with chronic neuromuscular disorders. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013170. doi: 10.1002/14651858.CD013170.pub2. PMID 33887060

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional Treatment | Lung Volume Recruitment
Started | 33 | 37
Completed | 28 | 25
Not Completed | 5 | 12
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 2 | 7
Not completed — Enrolled in drug trial | 3 | 1
Not completed — Became ineligible | 0 | 2

BASELINE CHARACTERISTICS:
Population: Of the 70 enrolled children, four did not have reliable or reproducible FVC measurements at baseline and were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Treatment | Lung Volume Recruitment | Total
Number analyzed (Participants) | 30 | 36 | 66
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 11.5 [9.2 to 13.0] | 11.5 [9.5 to 13.9] | 11.5 [9.5 to 13.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 36 | 66
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
FVC [Median (Inter-Quartile Range); unit: %-predicted] | 85.6 [73.8 to 98.8] | 84.0 [73.9 to 92.4] | 84.8 [73.3 to 95.5]
Wheelchair assisted [Count of Participants; unit: Participants] | 10 | 11 | 21
Scoliosis [Count of Participants; unit: Participants] | 3 | 6 | 9
Non-invasive ventilation [Count of Participants; unit: Participants] | 2 | 2 | 4
Steroid use [Count of Participants; unit: Participants] | 27 | 32 | 59

OUTCOME MEASURES:

1. Primary Outcome: Change in FVC (%-Predicted) From Baseline to 2 Years.
Description: Change in FVC (%-predicted) was chosen as the primary outcome as it is a strong predictor of subsequent respiratory failure and mortality. Although survival is not a realistic endpoint for this trial, given expected mortality is less than 5% for the pediatric age group, FVC change is an appropriate clinical laboratory measure and valid surrogate endpoint to use for this trial.
Time Frame: 2 years
Population: Of the 70 children randomized to a treatment arm, four children (n=3 in conventional treatment group; n=1 in LVR group) were excluded from the analyses as they did not have a reliable or reproducible pulmonary function test at baseline. All remaining children were included in the analyses except where no measurement was available.
Measure: Mean (Standard Deviation); unit: Mean difference in FVC %-predicted
Arm/Group | Conventional Treatment | Lung Volume Recruitment
Number analyzed (Participants) | 25 | 28
Mean difference in FVC %-predicted | -9.2 (17.3) | -6.4 (15.7)
Statistical Analysis 1: Comparison: Conventional Treatment vs Lung Volume Recruitment; Test type: Superiority; p = 0.68, ANCOVA — The a priori threshold for statistical significance was a two-sided p-value of 0.05; Mean Difference (Net) = 1.9, 95% CI 2-sided [-6.9 to 10.7] — The mean difference between the intervention and the control group in the change from baseline to 2 years was estimated. Estimates presented here are based on multiple imputation of missing values

2. Secondary Outcome: FVC Decline of 10% of Predicted
Description: The time to reach an FVC decline of 10% of predicted will be used to calculate a hazard ratio.
Time Frame: 2 years
Population: Of the 70 children randomized to a treatment arm, four children (n=3 in conventional treatment group; n=1 in LVR group) were excluded from the analyses as they did not have a reliable or reproducible pulmonary function test at baseline. All remaining children were included in the analyses.
Measure: Mean (Standard Error); unit: Months (restricted mean)
Arm/Group | Conventional Treatment | Lung Volume Recruitment
Number analyzed (Participants) | 30 | 36
Months (restricted mean) | 19.14 (1.59) | 21.70 (1.22)

3. Secondary Outcome: Number of Participants Prescribed Outpatient Oral Antibiotic Courses Between Baseline and 2 Years
Description: Total number of participants who received any antibiotic courses between baseline and two years
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Treatment | Lung Volume Recruitment
Number analyzed (Participants) | 30 | 36
Participants | 1 | 2

4. Secondary Outcome: Health-related Quality of Life From Baseline to 2 Years
Description: Measured biannually using the Pediatric Quality of Life Inventory (PedsQL 4.0). The PedsQL includes four subscales: Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning. Each subscale is scored from 0 to 100, with higher scores indicating better health-related quality of life. A total score is computed by averaging all subscale scores.
Time Frame: 2 years
Population: Participants who received either Conventional Treatment or Conventional Treatment plus LVR.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Conventional Treatment | Lung Volume Recruitment
Number analyzed (Participants) | 23 | 25
score on a scale | 2.0 [-7.8 to 6.8] | 3.8 [-4.8 to 11.1]

5. Secondary Outcome: Change in Difference Between Assisted and Unassisted Peak Cough Flow (PCF) From Baseline to 2 Years
Description: Change in the difference between assisted and unassisted peak cough flow (in liters per minute) from baseline to 2 years.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: PCF="liters per minute"
Arm/Group | Conventional Treatment | Lung Volume Recruitment
Number analyzed (Participants) | 2 | 3
PCF="liters per minute" | -2.6 (32.0) | 44.9 (65.6)
Statistical Analysis 1: Comparison: Conventional Treatment vs Lung Volume Recruitment; Difference in change in peak cough flow (L/min) from baseline to 2 years, between conventional treatment and intervention group; Test type: Superiority; Mean Difference (Net) = 0.27, 95% CI 2-sided [-1.92 to 2.18]

6. Secondary Outcome: Change in Maximal Insufflation Capacity (MIC)-Vital Capacity (VC) From Baseline to 2 Years
Description: Change in maximal insufflation capacity (MIC)-vital capacity (VC) in liters from Baseline to 2 Years
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: MIC-VC="Liter"
Arm/Group | Conventional Treatment | Lung Volume Recruitment
Number analyzed (Participants) | 7 | 9
MIC-VC="Liter" | 0.1 (0.2) | 0.0 (0.2)
Statistical Analysis 1: Comparison: Conventional Treatment vs Lung Volume Recruitment; Test type: Superiority; p = 0.79, Mixed Models Analysis

7. Secondary Outcome: Change in Maximum Inspiratory Pressures (MIP), From Baseline to 2 Years
Description: Change in maximum inspiratory pressures (MIP, in centimeters of water), From Baseline to 2 Years
Time Frame: 2 years
Population: Of the 70 children randomized, 4 (n=3 in conventional treatment group; n=1 in LVR group) were excluded from the analyses as they did not have a reliable or reproducible baseline pulmonary function tests. Results are for the observed population, as missing data imputation was not feasible. Of the remaining children, missing data was as follows: MIP and MEP (3 in conventional arm, 5 in LVR arm). A total of 16 children in the conventional group and 17 in the LVR group had useable data for MIP.
Measure: Mean (Standard Deviation); unit: "cm H2O"
Arm/Group | Conventional Treatment | Lung Volume Recruitment
Number analyzed (Participants) | 15 | 17
"cm H2O" | -0.5 (15.7) | -4.6 (25.1)
Statistical Analysis 1: Comparison: Conventional Treatment vs Lung Volume Recruitment; Test type: Superiority; p = 1.00, Mixed Models Analysis

8. Secondary Outcome: Change in Maximal Expiratory Pressures (MEP), From Baseline to 2 Years
Description: Change in maximal expiratory pressures (MEP, in liters), From Baseline to 2 Years
Time Frame: 2 years
Population: Of the 70 children randomized, 4 (n=3 in conventional treatment group; n=1 in LVR group) were excluded from the analyses as they did not have a reliable or reproducible baseline pulmonary function tests. Results are for the observed population, as missing data imputation was not feasible. Of the remaining children, missing data was as follows: MIP and MEP (3 in conventional arm, 5 in LVR arm). A total of 16 children in the conventional group and 17 in the LVR group had useable data for MEP.
Measure: Mean (Standard Deviation); unit: "cm H2O"
Arm/Group | Conventional Treatment | Lung Volume Recruitment
Number analyzed (Participants) | 16 | 17
"cm H2O" | 5.5 (17.1) | 12.9 (19.4)
Statistical Analysis 1: Comparison: Conventional Treatment vs Lung Volume Recruitment; Test type: Superiority; p = 0.98, Mixed Models Analysis

9. Other Pre Specified Outcome: Maximal and Average Pressure Achieved With LVR (cmH2O)
Time Frame: 2 years
Population: Data not collected during the study.
Arm/Group | Conventional Treatment | Lung Volume Recruitment
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Respiratory Symptoms
Description: Mean rate of symptom months over the study period. Symptom months are months with any respiratory symptom.
Time Frame: 2 years
Population: Respiratory symptoms were collected by telephone every 3 months over the study period.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Conventional Treatment | Lung Volume Recruitment
Number analyzed (Participants) | 28 | 32
Months | 0.08 (0.14) | 0.12 (0.29)

ADVERSE EVENTS:
Time Frame: 2 years (baseline to last follow-up at 2 years).
Arm/Group | Conventional Treatment | Lung Volume Recruitment
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/36
Other Adverse Events (participants affected / at risk) | 0/30 | 3/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Treatment (N=30) | Lung Volume Recruitment (N=36)
Mild chest discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Discomfort associated with use of LVR
Syncopal episode (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Probably related to LVR

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT01999075/Prot_SAP_000.pdf